CLINICAL TRIAL: NCT03956212
Title: Inflammatory Proteins, Gene Polymorphisms, and Transcriptome Profiles in Patients With Erythema Migrans
Brief Title: Inflammatory Mediators in Erythema Migrans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana School of Medicine, Slovenia (Other)
Responsible Party: Principal Investigator, Daša Stupica, Principal Investigator, University Medical Centre Ljubljana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EM Doxy-2017
Record Dates: First submitted 2019-05-15; First posted 2019-05-20 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Erythema Migrans
Keywords: Lyme Borreliosis; Inflammation; Outcome
MeSH Terms: conditions — Glossitis, Benign Migratory; Lyme Disease; Inflammation | interventions — Doxycycline

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- erythema migrans patients treated with doxycycline (Experimental): adult patients with erythema migrans will be treated with oral doxycycline
  Interventions: Drug: Doxycycline 7 days; Drug: Doxycycline 14 days

INTERVENTIONS:
Drug: Doxycycline 7 days — Patient will be treated with doxycycline orally, 100 mg, bid, 7 days
Drug: Doxycycline 14 days — Patient will be treated with doxycycline orally, 100 mg, bid, 14 days

SUMMARY:
The main objective of this study is to characterize the inflammatory proteins, gene polymorphisms, and transcriptome profiles in patients with erythema migrans to gain better insight into pathogenesis of early Lyme borreliosis and to define new immune modulators that could serve as biomarkers of disease activity.

ELIGIBILITY:
Inclusion Criteria:

* erythema migrans in patients > 18 years

Exclusion Criteria:

* pregnancy or immunocompromising conditions
* taking antibiotic with antiborrelial activity within 10 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
inflammatory proteins in erythema migrans patients | up to 12 months follow-up
  The inflammatory immune profiles will be assessed using Luminex to measure the expression of cytokines and chemokines representative of innate and adaptive TH1, TH2, TH17, and B cell responses in serum and if available, skin, of patients during active infection and after treatment.

SECONDARY OUTCOMES:
gene polymorphisms in erythema migrans patients | at enrollment
  ImmunoChip single-nucleotide polymorphism array for dense genotyping of rheumtic disease-relevant genomic variants will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Daša Stupica, MD PhD, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Medical Center Ljubljana, Ljubljana, Slovenia